CLINICAL TRIAL: NCT02628639
Title: Using High-resolution Electroencephalography to Optimize the Evaluation of Awareness in Patients With Disorders of Consciousness
Brief Title: Optimizing the Evaluation of Awareness in Disorders of Consciousness
Acronym: CONPHIDENSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/482
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electroencephalography recording (Experimental): Cerebral measurements from high-density electroencephalography after the presentation of personalized stimulations
  Interventions: Device: high-density electroencephalography

INTERVENTIONS:
Device: high-density electroencephalography

SUMMARY:
The purpose of this study is to evaluate whether personalized stimulations can improve the detection of electrophysiological signs of awareness in patients with disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* patients in a vegetative state or a minimally conscious state
* agreement from families

Exclusion Criteria:

* patients with akinetic mutism or locked-in syndrome
* patients in a coma
* patients with damages in the inner or middle ear
* contraindication to a high-density electroencephalography exam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants showing differences of electrophysiological activity after personalized but not standard stimulation protocols | standard stimulations: 28 days after recruiting patients
  Depending of the personalized stimulation protocol, the differences of electrophysiological activity can the presence of event-related potentials (N100, mismatch negativity, P300, etc.) or alterations of neural oscillations.
  The personalized stimulation protocol will be chosen according to the families' feeling of a presence.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Aubry, MD, PhD, Principal Investigator — Service douleur - soins palliatifs

REFERENCES:
- [Background] Pazart L, Gabriel D, Cretin E, Aubry R. Neuroimaging for detecting covert awareness in patients with disorders of consciousness: reinforce the place of clinical feeling! Front Hum Neurosci. 2015 Feb 17;9:78. doi: 10.3389/fnhum.2015.00078. eCollection 2015. No abstract available. PMID 25741272
- [Background] Gabriel D, Henriques J, Comte A, Grigoryeva L, Ortega JP, Cretin E, Brunotte G, Haffen E, Moulin T, Aubry R, Pazart L. Substitute or complement? Defining the relative place of EEG and fMRI in the detection of voluntary brain reactions. Neuroscience. 2015 Apr 2;290:435-44. doi: 10.1016/j.neuroscience.2015.01.053. Epub 2015 Jan 30. PMID 25644421